CLINICAL TRIAL: NCT05054712
Title: Prevalence of Metabolic Liver Diseases in Patients With Type 1 Diabetes Mellitus: Non-alcoholic Fatty Liver Disease and Glycogenic Hepatopathy
Brief Title: Prevalence of Metabolic Liver Diseases in Patients With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: 21-E5
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Non-alcoholic Fatty Liver Disease; Glycogen Hepatopathy; Type 1 Diabetes; Liver Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 1; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) has been extensively studied in the context of type 2 diabetes mellitus (T2D) due to its higher prevalence and its association with obesity and syndrome metabolic, a well-established risk factor for NAFLD. Although several studies have reported the accumulation of liver fat in patients with type 1 diabetes mellitus (T1D), the prevalence, etiology, and the consequences of NAFLD in patients with T1D are poorly characterized, requiring more studies in this field. In addition, liver involvement at the metabolic level in patients with T1D raises the differential diagnosis between NAFLD and glycogen hepatopathy (GH), a rare complication associated with the poorly metabolic control of diabetes and probably underdiagnosed, since the ultrasound pattern is the same than the NAFLD. The investigators have designed a cross-sectional observational study with the objective of describing the prevalence of metabolic liver diseases (NAFLD and GH) in the population of patients with T1D in the healthcare area of Hospital del Mar and Hospital de Vilafranca, as well as studying the relationship of these pathologies with the degree of metabolic control, the presence of metabolic syndrome and the presence of micro and macrovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years.
* Diagnosed with T1D of at least 6 months of evolution.
* Patients who give their informed consent in writing.

Exclusion Criteria:

* Active alcoholism> 30 g / day in men and> 20 g / day in women.
* Known non-metabolic liver disease: alcoholic hepatitis, viral hepatitis from HBV infection and / or HCV, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, autoimmune hepatitis, hepatic granulomatous (tuberculosis, mycobacteria, histoplasmosis), hepatic lymphoma, primary neoplasia liver, liver metastasis.
* Active treatment with hepatotoxic drugs: amiodarone, isoniazid, rifampicin, sulfa drugs, tetracyclines, amoxycline / clavulanate, ketoconazole, methotrexate, valproic acid, trazodone, tamoxifen, methyldopa, reverse transcriptase inhibitors, chemotherapy, immunotherapy.
* Pregnant women.
* Acute decompensation of T1D (ketoacidosis) in the 3 months prior to inclusion. The inclusion after this period.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Descriptive observational study of prevalence (cross-sectional) in patients with T1D of the healthcare area of the Hospital del Mar and Hospital de Vilafranca (Barcelona).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence of metabolic liver diseases (NAFLD and GH) by different diagnostic approaches in the population of patients with T1D. | 2 years
  To describe the prevalence of metabolic liver diseases (NAFLD and GH) by different diagnostic approaches (levels of transaminases, liver ultrasound, liver MRI and, in selected cases, liver biopsy) in the population of patients with T1D in the healthcare area of Hospital del Mar and Hospital de Vilafranca.

SECONDARY OUTCOMES:
To study the relationship between metabolic liver diseases in patients with T1D and the degree of metabolic control of diabetes. | 2 years
To study the relationship between metabolic liver diseases in patients with T1D and the presence of metabolic syndrome. | 2 years
To study the relationship between metabolic liver diseases in patients with T1D and the presence of microvascular and macrovascular complications. | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Comarcal de l'Alt Penedès, Vilafranca del Penedès, Barcelona
  - Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No